CLINICAL TRIAL: NCT03186560
Title: A Single Centre Open Label Study Measuring Microcirculatory Flux Using Speckle Imaging Device, in Patients With Arterial, Mixed and Diabetic Foot Ulcers Using gekoTM Neuromuscular Electrostimulation (NMES)
Brief Title: Speckle Study: In Arterial, Mixed and Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FSK-Speckle-001
Record Dates: First submitted 2017-06-05; First posted 2017-06-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Leg Ulcer
Keywords: Leg ulcers and use of geko device
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Intervention Model Description: Geko device will be provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Arterial Leg Ulcer (Active Comparator): Defined as healing/non-healing Healing defined as reduction in wound area of greater than 20% over a 2-week period
  Interventions: Device: gekoTM
- Group B: Mixed Leg Ulcer (Active Comparator): only to be done once Arterial leg ulcers show change in flux ABPI of <0.8-0.6
  Interventions: Device: gekoTM
- Group C: Diabetic Foot Ulcer - neuropathic (Active Comparator): On clinical inspection present as neuropathic
  Interventions: Device: gekoTM
- Group D: Diabetic Foot Ulcer - neuroischemic (Active Comparator): On clinical inspection present as neuroischemic
  Interventions: Device: gekoTM

INTERVENTIONS:
Device: gekoTM — The geko™ W devices are small disposable, internally powered, neuromuscular stimulators that are applied externally to the leg. The W device has a fixed 27mA current. The devices are self-adhesive and are applied to the outer/posterior aspect of the knee. This positioning enables integral electrodes to apply a stimulus to the lateral popliteal nerve (often additionally termed the common peroneal) which branches from the sciatic nerve. This nerve controls the contraction of several muscles in the lower leg.

SUMMARY:
This is a single centre open label study measuring microcirculatory flux using Speckle imaging Device.

Microcirculation will be measured using laser speckle contrast imaging, at baseline and with the device active for 30 minutes in the wound, peri-wound and other point on the lower leg. The same procedure will be done on all the different patient groups.

Temperature variations can be assessed using Infrared Temperature Scanner (Exergen DermaTemp DT1001), a measurement will be taken at baseline, and then at 5 minutes interval during the 30 minutes activity of the device.

DETAILED DESCRIPTION:
The most common underlying etiologic factors responsible for chronic delayed healing among lower extremity wounds encountered in the outpatient clinic are chronic venous insufficiency (CVI), diabetic neuropathy, and arterial insufficiency (AI). One or more of these factors can be identified in more than 90% of chronic lower extremity ulcers, and treatment protocols have been designed to manage wounds of each type to maximize healing potential. It is important to remember that multiple factors may coexist in any individual patient with a chronic wound, complicating management and hindering the healing process. Recently, it has been reported that the neuroischemic diabetic foot ulcer is now more common than nonischemic neuropathic diabetic foot ulcers, as arterial insufficiency promoted by poorly controlled diabetes complicates already impaired healing present in patients with diabetes.

Chronic leg ulcers are painful, debilitating wounds that place a significant burden on the patient, their family, and healthcare resources. Treating leg ulcers can present a significant challenge to clinicians, who currently have a limited range of treatments at their disposal. The mainstay of treatment is compression bandaging, ambulation and elevation at rest. In patients with mobility deficits, or in those who are unable to tolerate compression bandaging, ulcers may deteriorate and never heal. Accordingly, there is a need for novel, alternative devices or strategies that can be used to complement or replace compression therapy.

Numerous pathophysiological and metabolic factors can affect wound healing and result in a poor outcome. They include local causes such as oedema, ischemia, tissue hypoxia, infection, necrosis and growth factor imbalance, as well as systemic causes including metabolic disease, nutritional status general perfusion disturbances and pre-existing illness. These factors alter the wound repair environment, impede healing and increase the risk of chronic wound development. All healing processes including, inflammatory cell influx, fibroblast migration, and collagen and extracellular matrix deposition, are delayed in this situation, leading to prolonged wound healing.

Any wound management should assist the healing process and optimise the patient's blood flow to the wound area4. An acute wound in a stable patient with normal blood flow should heal successfully. Anything that compromises tissue oxygen delivery, such as poor vascularisation, will impede healing. There is a strong scientific basis for oxygen treatment as prophylaxis against infection; to facilitate wound closure and to prevent amputation in wounded patients. Oxygen delivery is a critical element for the healing of wounds. Hypoxemia, caused by disrupted vasculature, is a key limiting factor against wound healing.

The link between compromised circulation and ulceration is well established and well described. Chronic venous insufficiency is a direct cause of ulceration.

Diabetic foot ulcer is a major complication of diabetes mellitus, and probably the major component of the diabetic foot. Diabetes mellitus is one such metabolic disorder that impedes the normal steps of the wound healing process. Many studies show a prolonged inflammatory phase in diabetic wounds, which causes a delay in the formation of mature granulation tissue and a parallel reduction in wound tensile strength.

Treatment of diabetic foot ulcers should include: blood sugar control, removing dead tissue from the wound, dressings, and removing pressure from the wound through techniques such as total contact casting. Surgery in some cases may improve outcomes. Hyperbaric oxygen therapy may also help but is expensive. It occurs in 15% of people with diabetes and precedes 84% of all diabetes-related lower-leg amputations.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to enter the study patients must meet the following criteria:

* Age ≥ 18 years
* Intact healthy skin at the site of device application
* Able to understand the Patient Information Sheet
* Willing and able to give informed consent
* Willing and able to follow the requirements of the protocol
* Specific inclusion criteria for the subgroups:

Group A: Arterial Leg Ulcer

* Defined as healing/non-healing Group B: Mixed Leg Ulcer (only to be done once Arterial leg ulcers show change in flux)
* ABPI of <0.8-0.6 Group C: Diabetic Foot Ulcer - neuropathic
* On clinical inspection present as neuropathic Group D: Diabetic Foot Ulcer - neuroischemic
* On clinical inspection present as neuroischemic

Exclusion Criteria:

Patients will not be admitted to the study if they meet any of the following exclusion criteria:

* Significant (not colonialization) Wound infection either acute or chronic??
* History of significant haematological disorders or DVT with the preceding six months
* Pregnant
* Pacemakers or implantable defibrillators
* Use of any other neuro-modulation device
* Current use of TENS in pelvic region, back or legs
* Use of investigational drug or device within the past 4 weeks that may interfere with this study
* Recent surgery that may affect the study (such as abdominopelvic, or lower limb) in the opinion of the investigator.
* Recent trauma to the lower limbs that will prevent stimulation of the leg with geko (non-responders)
* Size of leg incompatible with the geko™ device., i.e prevents device from stimulating the common peroneal nerve
* obesity (BMI > 35)
* Any medication deemed to be significant by the Investigator
* Specific exclusion criteria for different subgroups:

Group A: Arterial Leg Ulcer - Mixed leg ulcer, diabetic foot ulcer or diabetic foot ulcer with neuroischaemic element.

Group B: Mixed Leg Ulcer

- Arterial leg ulcer, diabetic foot ulcer or diabetic foot ulcer with neuroischaemic element.

Group C: Diabetic Foot Ulcer - Mixed leg ulcer, Arterial leg ulcer, or diabetic foot ulcer with neuroischaemic element.

Group D: Diabetic Foot Ulcer - neuroischemic

- Mixed leg ulcer, Arterial leg ulcer or diabetic foot ulcer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Microcirculatory flux in the lower limb of the different subgroups with geko device on. | 35 minutes
  Measurements of microcirculatory flux in the lower limb of the different subgroups with geko device on.

SECONDARY OUTCOMES:
Temperature variation | 35 minutes
  measurements of Temperature over same time period as speckle device using the Exergen DermaTemp model DT1001.
Adverse Events | 35 minutes
  study rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Bosanquet, Principal Investigator — Aneurin Bevan University Health Board
Locations (3):
- United Kingdom (3):
  - Glenfield Hospital, Leicester
  - Aneurin Bevan Local Health Board, Newport
  - Welsh wound Innovation Centre, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosanquet DC, Ivins N, Jones N, Harding KG. Microcirculatory Flux and Pulsatility in Arterial Leg Ulcers is Increased by Intermittent Neuromuscular Electrostimulation of the Common Peroneal Nerve. Ann Vasc Surg. 2021 Feb;71:308-314. doi: 10.1016/j.avsg.2020.07.030. Epub 2020 Aug 5. PMID 32768540